CLINICAL TRIAL: NCT07372105
Title: Validation of the French Version of the Smile Esthetics-Related Quality of Life (SERQoL) Questionnaire
Brief Title: Validation of the French Version of the SERQoL Questionnaire
Acronym: Periosmile1
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251033
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Smile; Smile Esthetics
Keywords: smile esthetics; life quality; SERQoL; psychometric validation; patient-reported outcomes
MeSH Terms: conditions — Smiling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to validate the French version of the Smile Esthetics-Related Quality of Life (SERQoL) questionnaire in adult patients recruited in two APH-HP dental departments. The study evaluates internal consistency, test-retest reliability, and construct validity of the questionnary. A total of 120 patients will be recruited from dental departments at two AP-HP hospitals.

DETAILED DESCRIPTION:
This psychometric validation study involves adult patients receiving their first consultation at AP-HP dental services. The SERQoL questionnaire will be completed twice (at baseline and after 15 days). Internal consistency (Cronbach's alpha), test-retest reliability (intraclass or Pearson correlation), and factor structure (confirmatory factor analysis) will be analyzed. No clinical intervention is involved, and participation will not alter standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients attending their first periodontal consultation at the oral medicine departments of Rothschild Hospital (AP-HP) or Charles Foix Hospital (AP-HP)
* Patients who speak and understand French well enough to read and understand the study information sheet.
* Patients who are informed and do not object to participating in the study

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients who are completely edentulous, whether the edentulism is compensated or not

  * Patients with multiple dental agenesis (more than 6 teeth), amelogenesis, or syndromic or non-syndromic dentinogenesis imperfecta
  * Patients with psychiatric illnesses that may impact body image, such as patients with anorexia-bulimia or body dysmorphic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients attending a first consultation in the dental department of Rothschild or Charles Foix hospitals (AP-HP). Participants must speak and understand French and have not opposed participation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Measure of the internal consistency by the Cronbach's alpha | Day 15
  Measure of the questionnaire internal consistency by the Cronbach's alpha
Measure of the test-retest reliability by the intraclass or Pearson correlation | Day 15
  Measure of the questionnaire test-retest reliability by the intraclass or Pearson correlation
Measure of the factor structure by the confirmatory factor analysis. | Day 15
  Measure of the questionnaire factor structure by the confirmatory factor analysis

SECONDARY OUTCOMES:
Average score measure by gender | Day 0
  Average questionnaire score measure by gender
Average score measure by age | Day 0
  Average questionnaire score measure by gender
Average score measure according to periodontal health status | Day 0
  Average questionnaire score measure according to periodontal health status

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Rotschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided